CLINICAL TRIAL: NCT07110792
Title: A Mindfulness-based Intervention to Reduce Stress and Improve Prosocial Skills for Health-care Students : a Translational RCT Integrating Clinical, Neuroimaging and Biomedical Outcomes
Brief Title: A Mindfulness-based Intervention to Reduce Stress and Improve Prosocial Skills for Health-care Students
Acronym: e-SMILE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Geneva, Switzerland (Other)
Collaborators: Geneva University Hospital, Geneva, Switzerland (Unknown); SNF Swiss National Foundation (Unknown)
Responsible Party: Principal Investigator, Camille Nemitz Piguet, MD, PhD, PD, University of Geneva, Switzerland
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 2021-02059
Record Dates: First submitted 2025-07-23; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Mental Health Issue
Keywords: perceived stress; prosocial skills; health students; mindfulness; compassion skills; psychological well-being; MBCT-L
MeSH Terms: conditions — Psychological Well-Being | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: The intervention is compared to a waiting list group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clinical arm (Experimental): In this arm, participants complete clinical questionnaires
  Interventions: Other: Mindfulness-based Cognitive Therapy for Life (MBCT-L)
- Neurobiological arm (Experimental): In this arm, participants complete either MRI and or blood sample
  Interventions: Other: Mindfulness-based Cognitive Therapy for Life (MBCT-L)

INTERVENTIONS:
Other: Mindfulness-based Cognitive Therapy for Life (MBCT-L) — The MBCT-L (Bernard, Cullen & Kuyken, 2017) intervention is an 8-week group intervention, comprising a pre-course orientation session, eight 2-hour sessions, and a half-day silent session.
  MBCT-L was delivered synchronously online. MBCT-L group were led by one MBCT-L instructor

SUMMARY:
We aim to study the clinical immediate and long-term efficacy of a web-delivered MBCT-L protocol targeting bachelor and master health-care students in Geneva, as well as to study the correlations of clinical, neuroimaging and biomedical effects of such an intervention.

Primary objective: To evaluate the immediate and long-term effect of MBCT-L on reducing perceived stress and improving pro-social skills for health-care students, compared to a control group.

Secondary objective: To evaluate the immediate and long-term effect of MBCT-L on trait mindfulness, compassion, global psychological well-being, sleep quality, anxiety, depression, satisfaction in studies and resilience, to broaden the clinical understanding of the impact of such an intervention.

DETAILED DESCRIPTION:
This study is led jointly by Prof. C. Nemitz-Piguet, Dr F. Jermann, and Prof. S. Rudaz, who serve as co-principal investigators.

This study is funded by the Swiss National Science Foundation (Grant number: 32003B_205111 / 1)

ELIGIBILITY:
Inclusion Criteria:

* Eligibility criteria were applied to recruit second, third- or fourth-year health students in Geneva, Switzerland, who were at least 18 years old, had some interest in mindfulness, were available for the duration of the study, and agreed on refraining from regular mindfulness practice until allocated to the MBCT-L group.

Exclusion Criteria:

* Students were excluded if they had a current depressive episode, post-traumatic stress disorder, psychotic disorder, or substance dependency as identified through the Mini international Neuropsychiatric Interview (MINI). All participants received oral and written information about the trial and signed the informed consent form prior to the beginning of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Work package 1 (WP1) - Perceived stress | T0: baseline T1: 3 months from T0 T2: 9 months from T0
  Perceived stress as measured by the Perceived Stress Scale (PSS; score range: 0 -56; a higher score indicates a higher perceived stress level)
Work package 1 (WP1) - Prosocial skills | T0: baseline T1: 3 months from T0 T2: 9 months from T0
  Prosocial skills as measured by the Prosocialness Scale for Adults (PBS; score range: 16-80; a higher score indicate a greater tendency towards prosocial behaviors).
Work package 2 (WP2) - Socio-affective Video Task with Resting State (SoVT-Rest) | T0: baseline T1: 3 months from T0 T2: 9 months from T0
  Cortico-limbic emotion regulation network reactivity to psychological stress as measured by functional MRI (fMRI) in response to the SOVT-Rest
Work package 2 (WP2) - Montreal Imaging Stress Task (MIST) | T0: baseline T1: 3 months from T0 T2: 9 months from T0
  Cortico-limbic emotion regulation network reactivity to psychological stress as measured by functional MRI (fMRI) in response to the MIST
Work package 3 (WP3) - Metabolic | T0: baseline T1: 3 months from T0 T2: 9 months from T0
  Metabolic constitutive profiles
Work package 3 (WP3) - Lipid | T0: baseline T1: 3 months from T0 T2: 9 months from T0
  Lipid signalling profiles

SECONDARY OUTCOMES:
WP1 - Trait mindfulness | T0: baseline T1: 3 months from T0 T2: 9 months from T0
  Questionnaire: Five Facets of Mindfulness Questionnaire (FFMQ); score range: 39-195.
  A higher score indicates a higher level of trait mindfulness
WP1 - Compassion | T0: baseline T1: 3 months after T0 T2: 9 months after T0
  Sussex-Oxford Compassion Scale; compassion for the self; score range: 20-120 ; compassion for others; score range: 20-120.
  A higher score indicates a greater level of compassion
WP1 - Psychological well-being | T0: baseline T1: 3 months from T0 T2: 9 months from T0
  Psychological well-being scale; score range 18-108. A higher score indicates a greater psychological well-being
WP1 - Insomnia | T0: baseline T1: 3 months from T0 T2: 9 months from T0
  Sleep condition indicator; score range: 0-32 A higher score corresponds to better sleep
WP1 - Anxiety and depression | T0: baseline T1: 3 months from T0 T2: 9 months from T0
  Hospital Anxiety and Depression Scale; score range: 0-21 for anxiety and 0-21 for depression subscale. Higher scores correspond to higher anxiety and depression
WP1 - Satisfaction with studies | T0: baseline T1: 3 months from T0 T2: 9 months from T0
  Scale of satisfaction with Studies; score range 5-35. A higher score indicates a greater degree of contentment with one's academic experience
WP1 - Resilience | T0: baseline T1: 3 months from T0 T2: 9 months from T0
  Brief Resilience Scale; score range: 6-30. A higher score indicates a higher level of resilience
WP2 - Grey matter volume and functional connectivity in cortico-limbic emotion regulation networks (sMRI) | T0: baseline T1: 3 months from T0 T2: 9 months from T0
  Grey matter volume and functional connectivity in cortico-limbic emotion regulation networks (sMRI)
WP2 - Resting State neuroimaging data | T0: baseline T1: 3 months from T0 T2: 9 months from T0
  Resting State neuroimaging data
WP3 - Cortisol | T0: baseline T1: 3 months from T0 T2: 9 months from T0
  Capillary and blood cortisol
WP3 - Oxytocine | T0: baseline T1: 3 months from T0 T2: 9 months from T0
  Oxytocine
WP3 - Stress and inflammatory markers | T0: baseline T1: 3 months from T0 T2: 9 months from T0
  Stress and inflammatory markers

CONTACTS AND LOCATIONS:
Locations (1):
- University of Geneva, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No